CLINICAL TRIAL: NCT04489160
Title: A Phase II Trial on the Safety and Efficacy of C1 Inhibitor for the Acute Management of Severe Traumatic Brain Injury
Brief Title: Complement Inhibition: Attacking the Overshooting Inflammation @Fter Traumatic Brain Injury
Acronym: CIAO@TBI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Netherlands Brain Foundation (Other); Takeda (Industry)
Responsible Party: Principal Investigator, wcpeul, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL7255105823
Record Dates: First submitted 2020-07-17; First posted 2020-07-28 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Traumatic Brain Injury; Trauma, Head
Keywords: Traumatic Brain Injury; C1-inhibitor; Neuroinflammation; Efficacy; Safety
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma; Angioedemas, Hereditary; Neuroinflammatory Diseases | interventions — SERPING1 protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- C1-inhibitor (Experimental): One dose 6000 IU C1-inhibitor intravenously
  Interventions: Drug: C1 Inhibitor, Human
- Placebo (Placebo Comparator): 0.9% saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: C1 Inhibitor, Human — 6000 IU C1-INH
  Other Names: Cinryze
  Arms: C1-inhibitor
Drug: Placebo — 0.9% saline
  Arms: Placebo

SUMMARY:
Severe Traumatic Brain Injury (s-TBI) is a major cause of death and disability across all ages. Besides the primary impact, the pathophysiologic process of major secondary brain damage consists of a neuroinflammation response that critically leads to irreversible brain damage in the first days after the trauma. A key catalyst in this inflammatory process is the complement system. Inhibiting the complement system is therefore considered to be a potentially important new treatment for TBI, as has been shown in animal studies. This trial aims to study the safety and efficacy of C1-inhibitor compared to placebo in TBI patients. By temporarily blocking the complement system we hypothesize limitation of secondary brain injury and more favourable clinical outcome for TBI patients due to a decrease in the posttraumatic neuroinflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* Age at admission ≥ 18 years and < 65 years;
* Clinical diagnosis of traumatic brain injury with GCS < 13 (with intracranial deviations);
* Catheter placement for monitoring and management of increased ICP for at least 24 hours;

Exclusion Criteria:

* A clear, non-traumatic cause of low GCS (e.g. toxic, cardial) on admission;
* Not expected to survive more than 24 hours after admission;
* Brain death on arrival in the participating centers;
* Severe pre-trauma disability, defined as being dependent on other people;
* Known prior history of sensibility to blood products or Cinryze;
* Patients with a history of hereditary angioedema;
* Patients with a history of thrombosis;
* Pregnant women.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Therapy Intensity Level (TIL) Scale | First four ICU days
  TIL differentiated for various treatment modalities aimed at prevention or control of raised Intracranial Pressure (ICP) and/or for CPP management (0 to 38 points)
Glasgow Outcome Scale Extended (GOSE) | At 6 months after trauma
  Functional outcome (minimum score = 1, maximum score = 8)
Complication rate | Up to 1 year
  Adverse and serious adverse events related possibly related to study medication

SECONDARY OUTCOMES:
Intracranial pressure (ICP) burden | First four ICU days
  Minutes of ICP>20 mm Hg
CT scan midline shift | Up to 1 year
  in mm
Mortality | Up to 1 year after trauma
Glasgow Outcome Scale Extended (GOSE) | At discharge (an average of 14 days), 3 and 12 months after trauma
  Functional outcome (minimum score = 1, maximum score = 8)
QoLiBri | At 3, 6 and 12 months after trauma
  Quality of Life
SF-36 | At 3, 6 and 12 months after trauma
  Health-related quality of life
EQ-5D-5L | At 6 and 12 months after trauma
  Health-related quality of life
ICU length of stay | Up to 1 year
  in days
Ventilator days | Up to 1 year
  in days
Hospital length of stay | Up to 1 year
  in days
Hospital disposition | Up to 1 year
  Discharged to home, rehabilitation or nursery home
UCH-L1 and GFAP biomarkers | Baseline (Before adminstration of investigational product ) and 6, 12, 24, 48, 72 and 96 hours after adminstration of investigational product
Complement activation | Baseline (Before adminstration of investigational product ) and 6, 12, 24, 48, 72 and 96 hours after adminstration of investigational product
  WIESLAB, C3b/C, C4b/C, C5b-9 ELISA assays, CH50/AC50
Coagulation cascade activation | Baseline (Before adminstration of investigational product ) and 6, 12, 24, 48, 72 and 96 hours after adminstration of investigational product
  PT, aPPT, PLT, D-dimer, fibrinogen
Inflammatory markers | Baseline (Before adminstration of investigational product ) and 6, 12, 24, 48, 72 and 96 hours after adminstration of investigational product
  TNF-alpha, intraleukins

CONTACTS AND LOCATIONS:
Overall Officials: Wilco Peul, MD, MPH, PhD, MBa, Principal Investigator — Leiden University Medical Center
Locations (3):
- Netherlands (3):
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Center, Rotterdam
  - Haaglanden Medisch Centrum, The Hague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fluiter K, Opperhuizen AL, Morgan BP, Baas F, Ramaglia V. Inhibition of the membrane attack complex of the complement system reduces secondary neuroaxonal loss and promotes neurologic recovery after traumatic brain injury in mice. J Immunol. 2014 Mar 1;192(5):2339-48. doi: 10.4049/jimmunol.1302793. Epub 2014 Jan 31. PMID 24489093
- [Derived] van Erp IAM, van Essen TA, Fluiter K, van Zwet E, van Vliet P, Baas F, Haitsma I, Verbaan D, Coert B, de Ruiter GCW, Moojen WA, van der Jagt M, Peul WC. Safety and efficacy of C1-inhibitor in traumatic brain injury (CIAO@TBI): study protocol for a randomized, placebo-controlled, multi-center trial. Trials. 2021 Dec 4;22(1):874. doi: 10.1186/s13063-021-05833-1. PMID 34863258